CLINICAL TRIAL: NCT04899518
Title: A Phase 2b/3, Randomized, Double-Masked, Vehicle-Controlled Study Evaluating the Safety and Efficacy of Two Concentrations (0.4% and 1%) of ALY688 Ophthalmic Solution in Subjects With Dry Eye Disease (OASIS-1)
Brief Title: ALY688 Ophthalmic Solution in Subjects With Dry Eye Disease
Acronym: OASIS-1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Allysta Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALY688-301
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vehicle Ophthalmic Solution (Placebo Comparator)
  Interventions: Drug: ALY688 Ophthalmic Solution
- ALY688 Ophthalmic Solution Concentration 1 (Experimental)
  Interventions: Drug: ALY688 Ophthalmic Solution
- ALY688 Ophthalmic Solution Concentration 2 (Experimental)
  Interventions: Drug: ALY688 Ophthalmic Solution

INTERVENTIONS:
Drug: ALY688 Ophthalmic Solution — Ophthalmic Solution

SUMMARY:
Study Evaluating the Safety and Efficacy of Two Concentrations (0.4% and 1%) of ALY688 Ophthalmic Solution in Subjects with Dry Eye Disease

DETAILED DESCRIPTION:
Randomized, Double-Masked, Vehicle-Controlled Study Evaluating the Safety and Efficacy of Two Concentrations (0.4% and 1%) of ALY688 Ophthalmic Solution in Subjects with Dry Eye Disease

ELIGIBILITY:
Inclusion Criteria:

* Dry eye disease for > 3 months meeting specific sign and symptom criteria
* Best corrected visual acuity of +0.6 logMAR or better
* Willing to sign informed consent and attend study visits
* Willing to comply with contraception requirements

Exclusion Criteria:

* Unable to meet specific sign and symptom criteria
* Signs of ophthalmic allergic, inflammatory or infection conditions
* Use of contact lenses
* Anatomic abnormalities preventing accurate study assessments
* Use of medications that influence eye dryness
* Recent ophthalmic surgery
* Unwilling to suspend current treatments for dry eye disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 922 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Corneal fluorescein staining | 8 weeks
  Difference between ALY688 Ophthalmic Solution 0.4% and vehicle

CONTACTS AND LOCATIONS:
Locations (1):
- Allysta Pharmaceuticals, Bellevue, Washington, United States

IPD SHARING:
Plan to Share IPD: No